CLINICAL TRIAL: NCT00452231
Title: Comparative Study of the Efficacy of a Cognitive-Behavioral Therapy for Post-Traumatic Stress Disorder With or Without D-Cycloserine
Brief Title: RCT of CBT Combined With D-Cycloserine for Treating PTSD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Montréal (Other)
Collaborators: Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CRFS2045
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2007-03-27 (Estimated); Status verified 2007-03

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Post-traumatic Stress Disorder; Cognitive-Behavioral Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cycloserine; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: D-cycloserine
Behavioral: Cognitive-Behavioral Therapy

SUMMARY:
The purpose of this study is to investigate if the effectiveness of cognitive-behavioral therapy for post-traumatic stress disorder can be increased by combining it with D-cycloserine (TCC/D-cycloserine) by comparing with a placebo (TCC/placebo).

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is one of the most frequent anxiety disorder in the general population (Kessler and al., 2005). Currently, the treatment of choice for PTSD is cognitive-behavioral therapy (CBT; Foa, Davidson and Frances, 1999). Based on remission rates after treatment, successful outcomes of CBT for PTSD vary between 46 and 54 % when dropouts are considered, and between 56 and 70% among those who completed their therapy (Bradley and al., 2005). Thus, there is room for improvement.

Recently, the results of two published studies on the treatment of phobia of heights (Ressler and al., 2004) and social phobia (Hofman, 2006) indicated that the efficacy of CBT was increased by adding D-cycloserine. The superior efficacy of CBT/D-cycloserine over CBT/Placebo in the treatment of anxiety disorders can result from a greater release of glutamate, a substance facilitating the extinction of fear (Davis, Myers, Ressler and Rothbaum, 2005; Richardson, Ledgerwood an Cranney, 2004). However, to our knowledge, no study has yet compared CBT/D-cycloserine to CBT/Placebo in the treatment of PTSD. The main hypothesis of the current study is that the efficacy of CBT for PTSD will be increased when combined with D-cycloserine compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PTSD
* No other Axix I disorder of higher intensity than PTSD
* Accept not to start a psychopharmacological treatment before and during the participation to the project

Exclusion Criteria:

* Substance abuse
* Psychotic episodes (past or current)
* Bipolar disorder
* Organic caused mental disorder
* Intellectual deficiency
* Pregnant or breast-feeding woman
* Épilepsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2007-02; Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Clinician-administered measures collected at initial assessment, post-treatment and six-months follow-up:
CAPS: PTSD symptoms
SCID: AXIS I disorders

SECONDARY OUTCOMES:
Patient self-report forms collected at initial assessment, post-treatment and six-months follow-up:
BDI: depression symptoms
BAI: anxiety symptoms
WHOQL-Bref: quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Guay, Principal Investigator — Université de Montréal
Locations (1):
- Centre d'étude sur le Trauma, Montreal, Quebec, Canada